CLINICAL TRIAL: NCT00260143
Title: Testosterone and Physical Function in HIV Associate Weight Loss
Brief Title: Testosterone and Physical Function in HIV+ Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Charles Drew University of Medicine and Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: DK49296 (completed); CDU IRB#: 00-11-153-04 (Other: Charles R Drew University); R01DK049296 (NIH)
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: HIV Associate Weight Loss
Keywords: HIV+ men; Treatment Experienced
MeSH Terms: interventions — testosterone enanthate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Testosterone enanthate (Experimental): 300 mg of testosterone enanthate by intramuscular injection once weekly for 16 weeks
  Interventions: Drug: Testosterone enanthate
- Placebo (Placebo Comparator): Placebo (sesame oil) by intramuscular injection once weekly for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone enanthate
  Arms: Testosterone enanthate
Drug: Placebo
  Arms: Placebo

SUMMARY:
Men infected with the HIV virus (the virus that causes AIDS) often lose weight even though they may try to eat more food to gain weight. The reasons for this weight loss are not clear. Many men with HIV have low levels of testosterone in their blood. Testosterone is a hormone that is naturally produced in the bodies of both men and women and has important effects on building muscle and bone mass. The purpose of this study is to find out if providing additional testosterone to HIV infected men who have low testosterone can help them gain weight, increase their muscle mass, and feel better. The study will also help see if testosterone improves the efficiency with which your body produces and uses energy including fat. The dose of testosterone being used in this study will raise testosterone levels in the blood to higher than normal levels (2-3 times normal level).

DETAILED DESCRIPTION:
Purpose. Although the prevalence of weight loss in HIV-infected individuals has decreased in the developed world with the availability of highly active antiretroviral therapy, it continues to be a significant problem worldwide, and in the USA. The pathophysiology of weight loss in HIV-infected individuals is undoubtedly complex; decreased energy intake, metabolic dysregulation, intercurrent opportunistic infections, gastrointestinal infections and malabsorption, and hormonal abnormalities all contribute to the multifactorial origin of weight loss. Although patients with HIV-infection may lose both fat and lean tissue, the loss of lean body mass is an important aspect of the weight loss associated with wasting. Weight loss in HIV-infected patients is a good predictor of survival, risk of hospitalization, and opportunistic infections. The magnitude of depletion of nonfat tissues is an important determinant of the time of death in AIDS. One correctable factor in the complex pathophysiology of sarcopenia in HIV-infection is androgen deficiency. There is a high prevalence of low testosterone levels in HIV-infected men. Spontaneous and experimentally-induced androgen-deficiency in young men is associated with decreased muscle mass and strength. Testosterone replacement increases lean body mass, muscle strength, and muscle protein synthesis in androgen-deficient, young men. The studies supported by this grant in the previous budget period and others have demonstrated that testosterone replacement of HIV-infected men with weight loss and low testosterone levels is associated with an increase in fat-free mass and maximal voluntary muscle strength. Similarly, testosterone replacement of older men with low testosterone levels is associated with gains in fat-free mass and grip strength. However, it remains unknown whether testosterone-induced increases in fat-free mass and maximal voluntary strength are associated with clinically meaningful improvements in physical function and perceptions of physical function. Therefore, the primary objective of this competing renewal application is to determine if testosterone replacement of HIV-infected men with weight loss and low testosterone levels will improve objective measures of physical function, perceptions of physical function and body image. Our previous study demonstrated that testosterone replacement in HIV-infected men with low testosterone levels is associated with an increase in maximal muscle strength. However, testosterone effects on other important measures of muscle performance, such as power and fatigability that are important determinants of physical function, are not known. A second objective is to determine if testosterone replacement improves lower extremity power and fatigability.

The mechanisms by which testosterone increases muscle mass also remain unknown. Therefore, a third objective is to elucidate the mechanisms by which testosterone increases muscle mass and to determine its effects on energy balance.

Design. The study will be a randomized, placebo-controlled, double-blind study of HIV-infected men.

Sample Size Estimate. We estimate that approximately 50 men will be needed in each treatment group to test the proposed hypotheses (total 100 subjects).

Location: Subjects will be seen at the King/Drew Medical Center CRC (1720 E. 120th Street, Los Angeles, CA 90059) for all their visits.

Randomization and Subject Assignment. Subjects who meet the eligibility criteria will be randomly assigned to receive either testosterone enanthate (300 mg/weekly intramuscularly) or placebo.

Experimental Protocol. The study will consist of a screening phase, a 2-week control period, a 16-week treatment phase, and a 4-month recovery phase. We have selected a 16-week treatment period because the effects of testosterone on fat-free mass and muscle strength become manifest within this time period in healthy hypogonadal men, eugonadal men, and in HIV-infected men with weight loss.

Inclusion criteria A. Is the subject HIV positive, male and 18-60 years?

B. Is the subject wasting:

• a progressive weight loss within the previous 6 months of between 5-15 % of body weight, calculated by the equation (a-b)/a x 100% (a=highest weight in last6 months and b= present weight at screening), or • a BMI between 17 and 20 (= an actual body weight at screening of 85-95% of the lower limit of ideal weight), C. Is there an energy intake of calories of at least 80% of the estimated energy requirements? D. Is the subject On stable and potent antiretroviral therapy for at least 12 weeks, and in whom, in the opinion of the primary care provider, a change in antiretroviral therapy is unlikely in the next 4 months. Stable therapy may include those not on any antiretroviral therapies and whom, in the opinion of the primary care provider, will not be starting antiretroviral therapy in the next 4 months, E. Does the subject have a CD4 cell count > 50/mm3 or a viral load (HIV- copy number) < 10,000/ml ? F. Is the subject able and willing to comply with the trial protocol ? G. Is the subjects testosterone levels <400ng/dL? H. Is the subject able and willing to give informed consent in writing ?

Exclusion criteria

A. Does the subject have concurrent severe lipodystrophy according to the subject and the investigator? B. Does the subject have a history of hypersensitivity to anabolic steroids or to growth hormone? C. Does the subject have a history of prostatic or mammary cancer? D. Did the subject use nandrolone decanoate, growth hormone, androgen treatment or any other anabolic or appetite stimulating agents with the past 6 months ? E. Did the subject chronically use systematic corticosteroids (at least one month in the previous 6 months) except for topical applications? F. Does the subject have significant cardiac, renal, hepatic or other diseases that, in the opinion of the Investigator, may put the subject at risk if entered onto the trial or prevent successful completion of the trial ? 15. Has the subject had an AIDS defining illness (CDC HIV Classification, 1993: Clinical Category C)within the previous 3 months (except HIV wasting syndrome) ? G. Does the subject have a malignancy, other that Kaposi's Sarcoma localized to the skin ? H. Has the subject been involved in vigorous resistance exercise training programs (body building)in the last 3 months? 18. Dose the subject have diabetes mellitus? I. Is the active drug and/or alcohol use which would interfere with compliance for the study according to the investigator ? J. Did the subject receive investigational treatment except stable antiretroviral investigational drug in the last 12 weeks ?

K. Has the subject any of the following blood tests results:

Liver function test (ALAT/SGPT, ASAT/SCOT) > 5x the upper limit of the normal range (ULN) Cholesterol total > 3x ULN Alkaline Phosphotase >5 ULN or > 3xULN if bilirubin is above normal Serum Creatine > 2x ULN Platelet count < 50x 109 /L Haemoglobin < 8.0 g/L > 18g/dL PSA > 4 ng/ml Hct > 48 % L. Concomitant meds as exclusion (rhGh, IGF-1, other anabolic agents, appetite simulants, testosterone, ketoconazole, dilantin, phenobarbital, creatin, high dose of amino-acid supplements, protein supplements, androstenedione, DHEA & marinol)? M. Severe symptoms of BPH (American Urological Association [AUA] symptom index score of >14),prostate nodule, or induration on digital rectal examination [DRE] unless there has been a negative trans-rectal biopsy with last 3 months)? N. Untreated severe obstructive sleep apnea, as assessed by Berlin Symptom score? O. Limited neuromuscular, joint or some disease, or history of stroke with residual neurological defect that would preclude measurements of muscle strength of physical function? P. Significant diarrhea defined as 6 or more stools per day with recent change in bowel habits towards more frequent stools, especially if associated with weight loss and fever.

Outcome Measures

Our primary outcome measure is change from baseline in three important measures of physical function (stair climbing power, walking speed, and lifting task). These measures were selected because they are important for activities of daily living.

We will measure changes in maximal voluntary muscle strength, power, and muscle fatigability using the leg press exercise. This exercise was selected because it utilizes large muscle groups of the lower extremity that are important for functional activities, and is androgen-responsive (39).

Change in fat-free mass by dual energy X-ray absorptiometry (DEXA). Previous studies have already established that testosterone replacement increases fat-free mass. This study is focused on measures of muscle performance and physical function; therefore, we have not included more detailed assessment of body composition by deuterium water and sodium bromide.

Muscle volume of the non-dominant thigh will be measured by magnetic resonance imaging.

Intramuscular concentrations of myostatin, IGF-I, and IGFBP-4 mRNA will be measured by RT-PCR and protein by western blot analysis. The ubiquitin, and C3 and C9 proteasome mRNA will be measured by northern analysis.

Changes in perceptions of physical function, and body image. In addition to using global health related quality of life instruments, which have many domains that are not androgen-responsive, we will focus on assessment of perceptions of physical function, fatigue, and body image. These instruments have been demonstrated to be responsive to androgen replacement in older men with low testosterone levels (48).

Total and free testosterone, and dihydrotestosterone levels will be measured as markers of testosterone bioavailability. Serum LH, FSH and SHBG levels will be measured as markers of androgen action.

Safety Measures. Plasma lipids, apolipoproteins, and lipoprotein particles will be measured to assess testosterone effects on these markers of cardiovascular risk profile. Hemoglobin, liver enzymes (ALT, AST, bilirubin, GGT, alkaline phosphatase), serum PSA, digital rectal examination and AUA BPH symptom score will be monitored as safety parameters.

Energy Expenditure.. We will measure resting energy expenditure by indirect calorimetry, using a novel, handheld device known as the MedGem (HealtheTech, Golden Colorado) Neiman et al (Neiman DC, Trone GA, Austin MD. A new handheld device for measuring resting metabolic rate and oxygen consumption. J Am Diet Assoc 2003; 103(5 588-593) have validated this device in 63 males adult men and women with BMI between 19 and 56 kg/m2 against Douglas bags with duplicate measurements on each of two nonconsecutive days within a 14 day period. Since there were no differences between tests or between days for either the MedGem or the Douglas bags, the four tests for each device were pooled. The mean difference for the pooled results between MedGem and Douglas bags was 7 Kcal/day (0.4%). The thermic effect of food will be measured by indirect calorimetry, using the same MedGem apparatus with measurements during the last 15 minutes of each of five hours after ingestion of a standardized meal. We will also measure resting energy expenditure by use of the Deltatrac II device. After subjects have rested in bed for at least 5 minutes, oxygen consumption and carbon dioxide production will be measured using a ventilated canopy system for 20 minutes (Deltatrac II).

The rates of ATP synthesis will be measured by 31P and 13C nuclear magnetic resonance (NMR) spectroscopy. The rates of substrate oxidation in the citric acid cycle will be estimated from the specific activity of 4-13C glutamate during steady state infusion of 13C-1 acetate. The ratio of ATP synthesis measured by NMR spectroscopy and fuel oxidation measured by steady state 13-1 acetate infusion will be used as a measure of mitochondrial coupling of oxidation and phosphorylation. In addition, we will also measure mitochondrial energy coupling in isolated muscle fibers obtained from biopsies of vastus lateralis directly by measuring P:O ration using an oxygen electrode.

Body core temperature will be measured by obtaining rectal temperature, using a precise and accurate thermo-couple thermister.

Free fatty acid flux and adipose tissue lipolysis will be measured using [1-13C] palmitate and[2H5] glycerol isotope infusion, respectively. Fat oxidation will be measured by the release and quantitation of 1-13C-CO2 released during exhalation after infusion of the [1-13C] palmitate. [2H2] glucose isotope will be used to measure insulin sensitivity. One to two weeks before the second palmitate infusion, a single injection of sodium [1-13C] bicarbonate (1.76 µmol/kg; 90% enriched, sterile and pyrogen free; Mass Trace) will be used to calculate the acetate correction factor (ACF). The ACF accounts for 13C-label lost in exchange reactions in the tricarboxylic acid cycle. After 135 min of tracer equilibration, breath samples will be obtained in 15-min intervals up to 150 minutes and 5 minute intervals from 150 to 180 minutes. Non-esterified free fatty acid levels will be measured at baseline, mid-study (day 56) and at the end of treatment by a fasting blood measurement.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive men, 18-60 years of age, with objective evidence of HIV-infection with low to low-normal testosterone levels (<400 ng/dL). In boys before the age of 18, the hormonal and body composition changes of puberty can confound the data. We will exclude men over 60 because of age-related changes in testosterone levels and body composition, and increased risk of prostate disease.
* Documented weight loss within the previous 6 months of between 5-15% of body weight, or an actual body mass index (BMI) at screening of between 17 and 20 (= 85-95% of the lower limit of ideal weight).
* An energy intake of at least 80% of the estimated requirements. On stable and potent antiretroviral therapy for at least 12 weeks, and in whom, in the opinion of the primary care provider, a change in antiretroviral therapy is unlikely in the next 4 months. Stable therapy may include those not on any antiretroviral therapies and whom, in the opinion of the primary care provider, will not be starting antiretroviral therapy in the next 4 months CD4 cell count >50 /mm3, and HIV-copy number less than 10,000 copies/ml Testosterone levels <400ng/dL Able and willing to provide informed consent and comply with the protocol

Exclusion Criteria:

* Concurrent severe lipodystrophy* according to the patient and the investigator, defined as "the new appearance of thin extremities due to loss of subcutaneous fat (especially the medial compartment of the thigh) along with the new appearance of prominent veins. Loss of tissue in the buccal fat pad and subgluteal region provides further evidence that thin extremities may be in large part due to loss of fat and not just muscles."
* History of prostatic or mammary cancer
* Significant diarrhea defined as 6 or more stools per day with recent change in bowel habits towards more frequent stools, especially if associated with weight loss and fever
* Use of any androgen, growth hormone, or other anabolic or orexigenic agents within the past 6 months
* Use of systemic corticosteroids, except for topical application
* Significant cardiac, renal, hepatic or other diseases that, in the opinion of the Investigator, may put the subject at risk if entered onto the trial or prevent successful completion of the trial.
* AIDS defining illness (CDC HIV Classification, 1993: Clinical Category C) within the previous 3 months (except HIV wasting syndrome)
* Malignancy, other than Kaposi's Sarcoma localized to the skin
* Involvement in (vigorous) resistance exercise training programs (body building) in the past 3 months
* Diabetes mellitus Limiting neuromuscular, joint or bone disease, or history of stroke with residual neurological defect that would preclude measurements of muscle strength or physical function
* Severe symptoms of BPH (American Urological Association [AUA] symptom index score of >14), prostate nodule or induration on digital rectal examination (DRE) unless there has been a negative transrectal biopsy within 3 months, and prostate specific antigen (PSA) > 4
* Untreated severe obstructive sleep apnea, as assessed by Berlin's symptom score.
* Current alcohol or drug dependence which would interfere with compliance for the study
* Subject receive investigational treatment except stable antiretroviral investigational drug in the last 12 weeks
* Subject have a history of hypersensitivity to anabolic steroids or to growth hormone
* Any of the following blood test results:

  * Liver function test (ALT, AST) 5x the upper limit of the normal range (ULN)
  * Alkaline Phosphotase > 5x ULN or > 3x ULN if bilirubin is above normal
  * Cholesterol total (> 5 x ULN) or triglycerides 700 mg/dL
  * Serum Creatinine 2x ULN
  * Hemoglobin 8.0 g/dl or >18 g/dL
  * Platelet count < 50x109/L
  * HCT >48%
  * PSA 4 ng/ml.
* Concomitant Medications: Men who have received in the preceding 6 months or are currently using androgenic steroids, rhGH, IGF-I or other anabolic agents or appetite stimulants will be excluded. Also, excluded are drugs that affect testosterone secretion or metabolism such as ketoconazole, dilantin, and phenobarbital. Patients who have been on a stable dose of erythropoietin for at least 3 months will be allowed to continue the drug. The changes in antiretroviral therapy except for changes within the same class of drugs are not allowed. The use of corticosteroids, except for topical application, is not allowed. The food supplements that might affect body composition such as creatine, high dose amino-acid supplements, whey protein supplements, androstenedione, DHEA, and marinol, are also not allowed.
* On the Exclusion of Women. Women are not being included in this study because testosterone administration in these doses will inevitably cause virilization, and is ethically unacceptable.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2003-05 (Actual); Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Stair climb | 16 weeks
  A modification of the Margaria stair climb was used to assess stair-climbing power. participants were instructed to ascend a 12-step staircase as rapidly as possible, with ascent time recorded over the middle four steps (0.66 m) of the climb.
Walking speed | 16 weeks
  Participants were instructed to walk a 160-m flat course as fast as possible without running. Photoelectric cells and timers were used to determine time to the nearest 0.01 s. The faster of two trials was used to calculate walking speed (m/s).
Load carry | 16 weeks
  To simulate daily activities such as carrying groceries or suitcases, participants carried a load equal to 20% of their body weight while walking a distance of 20 m as fast as possible on a flat course.

CONTACTS AND LOCATIONS:
Overall Officials: Shalender Bhasin, MD, Principal Investigator — Charles R. Drew University and Boston University Medical Center
Locations (1):
- Charles R. Drew University, Los Angeles, California, United States

REFERENCES:
- [Result] Knapp PE, Storer TW, Herbst KL, Singh AB, Dzekov C, Dzekov J, LaValley M, Zhang A, Ulloor J, Bhasin S. Effects of a supraphysiological dose of testosterone on physical function, muscle performance, mood, and fatigue in men with HIV-associated weight loss. Am J Physiol Endocrinol Metab. 2008 Jun;294(6):E1135-43. doi: 10.1152/ajpendo.90213.2008. Epub 2008 Apr 22. PMID 18430965